CLINICAL TRIAL: NCT06145854
Title: Real World Clinical Outcomes in Cisgender Female Patients Who Start on Long Acting Cabotegravir for PrEP: An Observational, Multisite Prospective 2 Year Study in the Southern U.S.
Brief Title: Cisgender Female Patients Who Start on Long Acting Cabotegravir for PrEP
Status: Active, not recruiting | Type: Observational
Sponsor: Midway Specialty Care Center (Other)
Responsible Party: Principal Investigator, Emmanuelle Allseits, Physician, Midway Specialty Care Center
Other Study IDs: 2022-01
Record Dates: First submitted 2023-11-17; First posted 2023-11-24 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — cabotegravir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cisgender Females
  Interventions: Drug: Cabotegravir Injection [Apretude]

INTERVENTIONS:
Drug: Cabotegravir Injection [Apretude] — Apretude for PrEP

SUMMARY:
Oral PrEP regimens (FTC/TDF have been the mainstay of HIV prevention however patients now have more options for HIV prevention. In addition to oral PrEP regimens, the FDA approved the use of long acting Cabotegravir (CAB-LA) as the first long-acting medication for HIV prevention. This study will evaluate real world clinical outcomes of cisgender female patients who start CAB-LA for PrEP.

ELIGIBILITY:
Inclusion Criteria:

1. Cisgender females, ages 18 years and older
2. Negative HIV test at baseline
3. Negative Pregnancy test at baseline
4. Weigh at least 35 kilograms
5. Already Prescribed CAB-LA (Apretude)

Exclusion Criteria:

1. Transgender females or males
2. Cisgender males
3. Cisgender female who is actively breastfeeding
4. Severe hepatotoxicity
5. Evidence of Hepatitis B Infection
6. History or presence of allergies to cabotegravir or its components

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: 100 cisgender females (including 15 cisgender females with history of substance use and 15 cisgender females with unstable housing)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Describe the percent of cisgender females persistent on CAB-LA over 44 weeks. | 44 Weeks

SECONDARY OUTCOMES:
Describe incidence of bacterial STIs through weeks 20, 44 and 92 | Weeks 20, 44 and 92
Describe satisfaction of cisgender female patients while being on CAB-LA through weeks 20, 44 and 92 with the use of satisfaction surveys | Weeks 20, 44 and 92
Describe percentage adherence to CAB-LA injection schedule at weeks 20, 44 and 92 for cisgender females | Weeks 20, 44 and 92
Describe percentage adherence to CAB-LA injection schedule at weeks 20, 44 and 92 for cisgender females with substance use and/or unstable housing. | Weeks 20, 44 and 92
Describe percentage of cisgender female patients with HIV prevention failure while on CAB-LA, with detection of HIV, at weeks 20, 44 and 92. | Weeks 20, 44 and 92
Describe percentage of cisgender female patients with weight gain > 10% from baseline on CAB-LA at weeks 20, 44 and 92 | Weeks 20, 44 and 92

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Midway Specialty Care Center, Orlando, Florida
  - Midway Specialty Care Center, Temple Terrace, Florida
  - Midway Specialty Care Center, West Palm Beach, Florida

IPD SHARING:
Plan to Share IPD: No